CLINICAL TRIAL: NCT04743765
Title: HIP Fracture Accelerated Surgical TreaTment And Care tracK 2 (HIP ATTACK-2) Trial
Brief Title: HIP Fracture Accelerated Surgical TreaTment And Care tracK 2 Trial
Acronym: HIP ATTACK-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: v2.0_20230608
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hip Fractures; Myocardial Injury
MeSH Terms: conditions — Hip Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Accelerated medical clearance and surgery (Experimental): Accelerated medical clearance and targeted arrival to the operating room within 6 hours of eligibility criteria met.
  Interventions: Other: Accelerated medical clearance and surgery
- Standard surgical care (No Intervention): Hip fracture repair and surgical care according to treating institution guidelines.

INTERVENTIONS:
Other: Accelerated medical clearance and surgery — Rapid medical clearance with targeted arrival to the operating room within 6 hours of eligibility criteria criteria met.
  Arms: Accelerated medical clearance and surgery

SUMMARY:
The HIP ATTACK-2 trial is a multicentre, international, parallel group randomized controlled trial to determine whether accelerated surgery for hip fracture in patients with acute myocardial injury is superior to standard care in reducing death at 90 days after randomization. The trial will also assess secondary outcomes at 90 days after randomization: inability to independently walk 3 metres, time to first mobilization (first standing and first full weight bear), composite and individual assessment of major complications (e.g., mortality, non-fatal myocardial infarction, acute congestive heart failure, and stroke), delirium, length of stay, pain, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥45 years;
2. diagnosis of hip fracture during working hours with a low-energy mechanism requiring surgery;
3. troponin elevation ( at least one troponin measurement above the upper limit of normal occurring from the time of hip fracture to the time of randomization); and
4. informed consent.

Exclusion Criteria:

1. taking a therapeutic dose of an anticoagulant for which no reversing agent is available and the anesthesiologist or surgeon believe surgery within 6 hours of eligibility criteria met would not be safe;
2. patients on a therapeutic vitamin K antagonist with a history of heparin induced thrombocytopenia (HIT);
3. patients with peri-prosthetic fracture, open fracture or bilateral fractures;
4. patients requiring an emergency surgery for another reason (e.g., subdural hematoma);
5. patients with acute myocardial infarction deemed to be clinically unstable, with a mechanical complication (i.e., acute papillary muscle rupture, ventricular septal defect), ST elevation myocardial infarction, or cardiogenic shock;
6. patients refusing consent; or
7. patients previously enrolled in HIP ATTACK-2.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Within 90 days post randomization
  Death due to all causes

SECONDARY OUTCOMES:
Ability to independently walk 3 meters | Within 90 days post randomization
  Ability to independently walk 3 meters (10 feet) or across a room without human assistance. Patients who require a cane or walker, but not human assistance, will be classified as able to walk independently. Patients who require assistance to get out of a chair, but can walk independently once they get up, will be classified as able to walk independently.
Composite of major complications | Within 90 days post randomization
  Composite includes vascular and nonvascular mortality, non-fatal myocardial infarction, acute congestive heart failure, and stroke.
Vascular mortality | Within 90 days post randomization
  Any death with a vascular cause and includes those deaths following a myocardial infarction, sudden cardiac arrest, stroke, cardiac revascularization procedure (i.e., percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG] surgery), heart failure, pulmonary embolus, cardiovascular hemorrhage, or deaths due to an unknown cause
Nonvascular mortality | Within 90 days post randomization
  Any death due to a clearly documented non-vascular cause.
Myocardial Infarction | Within 90 days post randomization
  Diagnosis of MI according to 4th universal definition of myocardial infarction
Acute Congestive Heart Failure | Within 90 days post randomization
  at least one clinical sign(s) or symptom(s) (e.g elevated jugular venous pressure, respiratory rales/crackles, crepitations, hypoxia, tachypnea or presence of S3) with at least one of the following:
  1. radiographic findings (i.e., vascular redistribution, interstitial pulmonary edema, or frank alveolar pulmonary edema) or point of care ultrasound findings (i.e., bilateral B-lines, bilateral pleural effusion, elevated jugular venous pressure, dilated inferior vena cava with respiratory variation less than 50%) OR
  2. heart failure treatment implemented with diuretics with documented clinical improvement.
Stroke | Within 90 days post randomization
  Either - 1. a new focal neurological deficit thought to be vascular in origin with signs or symptoms lasting more than 24 hours or leading to death; or 2. a new focal neurological deficit thought to be vascular in origin with signs or symptoms lasting less 24 hours with a positive neuroimaging consistent with a stroke
Time from randomization to hospital discharge | Within 90 days post randomization
  Length of hospital stay from randomization to hospital discharge
Delirium | Within 7 days and 90 days post randomization
  1. Patient meets the criteria for delirium on any in-person 3D-CAM or CAM administered; OR
  2. Positive history of delirium in the 7 days after randomization based on the review of hospital health records.
Moderate to severe pain | Within 7 days and 90 days post randomization
  Moderate to severe pain is defined as any pain score ≥3 on 10 points scale.

OTHER OUTCOMES:
New clinically important atrial fibrillation or flutter | Within 90 days post randomization
  Documentation of atrial fibrillation or atrial flutter of any duration on an ECG, telemetry tracing, or rhythm strip and results in angina, congestive heart failure, symptomatic hypotension, or is followed by initiation or a dose increase of a rate controlling drug, antiarrhythmic drug, or electrical cardioversion.
Cardiac revascularization procedure | Within 90 days post randomization
  Revascularization procedures including coronary artery bypass graft or percutaneous coronary intervention surgery.
Venous thromboembolism | Within 90 days post randomization
  Venous pulmonary embolism or deep venous thrombosis
Pulmonary embolism | Within 90 days post randomization
  The diagnosis of PE requires any one of the following:
  1. A high probability ventilation/perfusion lung scan,
  2. An intraluminal filling defect of a segmental or larger artery on a helical CT scan,
  3. An intraluminal filling defect on pulmonary angiography, or
  4. A positive diagnostic test for DVT (e.g., positive compression ultrasound) and one of the following:
  A. Non-diagnostic (i.e., low or intermediate probability) ventilation/perfusion lung scan B. Non-diagnostic (i.e., subsegmental defects or technically inadequate study) helical CT scan.
Proximal deep venous thrombosis | Within 90 days post randomization
  The diagnosis of proximal DVT requires:
  1. Thrombosis involving the popliteal vein or more proximal veins for leg DVT and axillary or more proximal veins for arm DVT, AND
  2. Evidence of vein thrombosis by any one of the following:
  1. A persistent intraluminal filling defect on contrast venography, 2. Noncompressibility of one or more venous segments on B mode compression ultrasonography, or 3. A clearly defined intraluminal filling defect on contrast enhanced computed tomography.
Infection | Within 90 days post randomization
  Pathologic process caused by the invasion of normally sterile tissue or fluid or body cavity by pathogenic or potentially pathogenic organisms.
Sepsis | Within 90 days post randomization
  Based on the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) criteria,20 sepsis will require a quick Sequential Organ Failure Assessment (qSOFA) Score ≥2 points or patients requiring vasopressors/inotropes due to infection. The qSOFA includes the following items and scoring system:
  1. Altered mental status (1 point),
  2. Systolic blood pressure (SBP)of 100 mm Hg or less (1 point), and
  3. Respiratory rate (RR) of 22 breaths/min or more (1 point).
Pneumonia | Within 90 days post randomization
  Acute infection of the pulmonary parenchyma that is associated with at least one sign or symptom of lower respiratory acute infection (e.g., cough, pleuritic chest pain) or acute systemic illness (e.g., fever, chills, confusion, hypoxemia); accompanied by the presence of an acute infiltrate/consolidation on a chest radiograph or auscultatory findings consistent with pneumonia (such as crackles and/or localized rales) for which there is no other explanation.
Bleeding | Within 90 days post randomization
  Life threatening, major or critical organ bleeding
Hip reoperation | Within 90 days post randomization
  Any second surgical procedure undertaken on the fractured hip being followed in the study, for any reason (e.g. infection, implant failure, periprosthetic fracture, wound dehiscence, etc.), after it has been initially repaired and the patient has left the operating room.
Prosthetic hip dislocation | Within 90 days post randomization
  Any acute dislocation of a prosthetic femoral head from within its intended concentric location within the acetabulum. The acetabulum may or may not be resurfaced/replaced.
Implant failure | Within 90 days post randomization
  Any mechanical issue related to the integrity of any component of the hip implant which requires a surgical procedure to correct. This includes: loss of implant fixation to bone (either with or without associated periprosthetic fracture); or broken, disassociated, or dislocated implant components.
Peri-prosthetic fracture | Within 90 days post randomization
  Fracture through any part of either the femur and/or acetabulum to which a hip implant used for hip repair/reconstruction was fixed.
Acute kidney injury | Within 90 days post randomization
  An increase in the serum creatinine concentration from the pre-randomization value of ≥26.5 μmol/L (≥0.3 mg/dL) within 48 hours after randomization, or an increase of ≥50% within 7 days after randomization.
Acute renal failure resulting in dialysis | Within 90 days post randomization
  New requirement for dialysis (i.e., use of hemodialysis machine or peritoneal dialysis apparatus in patients without a requirement for dialysis prior to randomization).
Hospital re-admission | Within 90 days post randomization
  Hospital re-admission following discharge from index hospitalization
Length of critical care stay | Within 90 days post randomization
  Length of critical care stay
Length of rehabilitation stay | Within 90 days post randomization
  Length of rehabilitation stay
Days alive at home | Within 90 days post randomization
  Days alive at home are the number of days patients spend at their usual residence without, during that day, being admitted to a hospital or visiting an emergency department or urgent-care centre. Patients lose days alive at home if 1. patients go to an emergency department or urgent-care centre; 2. they become inpatients at a hospital or rehabilitation or convalescence-care facility; or 3. they die.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Borges, M.D, Principal Investigator — Population Health Research Institute; Gerard Slobogean, M.D, Principal Investigator — University of Maryland, Baltimore; Robert Feibel, M.D, Principal Investigator — The Ottawa Hospital; PJ Devereaux, M.D, Study Chair — Population Health Research Institute
Locations (70):
- United States (19):
  - Chandler Regional Medical Center, Chandler, Arizona
  - The Regents of the University of California, Davis, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Emory University at Grady Memorial Hospital, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Bryan Medical Center, Lincoln, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- The John Hunter Hospital, New Lambton Heights, New South Wales, Australia
- Cliniques Universitaires Saint Luc - University Catholic of Louvain, Woluwe-Saint-Lambert, Brussels Capital, Belgium
- University of São Paulo, São Paulo, São Paulo, Brazil
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - Victoria Hospital, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - CISSS de Laval, Laval, Quebec
- Chile (2):
  - Pontifica Universidad Catolica de Chile, Santiago, RM
  - Clinica Santa Maria, Santiago
- Finland (2):
  - South Karelia Central Hospital, Lappeenranta
  - Tampere University Hospital, Tampere
- Queen Mary Hospital, Hong Kong, Hong Kong
- India (5):
  - Bangalore Baptist Hospital, Bangalore, Karnataka
  - Government TD Medical College, Alappuzha, Kerala
  - Government Medical College, Trivandrum, Kerala
  - All India Institute of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - JIPMER, Puducherry, Puducherry
- Italy (4):
  - Hospital of Perugia, Perugia, Umbria
  - Galliera Hospital, Genova
  - Ospedale San Raffaele S.r.l., Milan
  - Ospedale Galeazzi SpA, Milan
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia
- Mexico (2):
  - Christus Muguerza del Parque, Chihuahua City, Chihuahua
  - Cruz Verde Guadalajara, Guadalajara, Jalisco
- B and B Hospital, Lalitpur, Bagmati, Nepal
- Netherlands (2):
  - Deventer Hospital, Deventer, Overijssel
  - Stichting OLVG, Amsterdam
- Pakistan (7):
  - Maroof International Hospital, Islamabad, ICT
  - Shifa International Hospitals Ltd., Islamabad, ICT
  - Hayat Abad Medical Complex, Peshawar, KPK
  - Ghurki Trust Teaching Hospital, Lahore, Punjab Province
  - Combined Military Hospital, Rawalpindi, Punjab Province
  - Aga Khan University, Karachi, Sindh
  - Indus Hospital & Health Network, Karachi, Sindh
- SPZOZ Myslenice, Myślenice, Malopolska, Poland
- King Faisal Specialist Hospital, Riyadh, Riyadh Region, Saudi Arabia
- South Africa (2):
  - Stellenbosch University - Tygerberg Hospital, Cape Town, Western Cape
  - Groote Schuur Hospital, Cape Town, Western Cape
- Spain (10):
  - Hospital Universitari Sagrat Cor, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic of Barcelona, Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona
  - Hospital Sant Camil, Sant Pere de Ribes, Barcelona
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Costa del Sol, Marbella, Malaga
  - Hospital Clinico Universitario de Vallad, Valladolid, Valladolid
  - Parc Sanitari Sant Joan de Déu, Barcelona

IPD SHARING:
Plan to Share IPD: No
The Population Health Research Institute (PHRI) is the sponsor of this trial. The PHRI believes the dissemination of clinical research results is vital and sharing of data is important. PHRI prioritizes access to data analyses to researchers who have worked on the trial for a significant duration, have played substantial roles, and have participated in raising the funds to conduct the trial. PHRI balances the length of the research study, and the intellectual and financial investments that made it possible with the need to allow wider access to the data collected. Data will be disclosed only upon request and approval of the proposed use of the data by a Review Committee.